CLINICAL TRIAL: NCT04261595
Title: Evaluating Dates as a Functional Food for Autism Via Its Prebiotic Effect, Modulation of Anti-Inflammatory and Anti-Oxidative Activity.
Brief Title: Dates as a Functional Food for Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Prof.Dr. Ammal Mokhtar Metwally, Principal Investigator, National Research Centre, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12060158
Record Dates: First submitted 2020-02-01; First posted 2020-02-10 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Autistic Spectrum Disorder
Keywords: Dates; Autism; microbiota; antioxidant; anti- inflammatory
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Functional Food; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Dates and their constituents show a role in disease prevention through anti-oxidant, anti-inflammatory, anti-bacterial activity. Dates are considered a staple food item in the Middle East and North Africa and are also imported in Europe, the UK, and the USA. (12).
  Dates' therapeutic effect in the management of the disease via its anti-oxidant, anti-inflammatory effect and for the sake of autistic children, is worthy to point and essential to evaluate Dates as a good remedy for autistic children because it is inexpensive and easy to access.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dates group 1 (Active Comparator): For the group of the date 1, Diagnosed autistic patients will be given three pieces of Dates will be given on daily basis for 12 weeks as follow: Three pieces (each about 10 -15 gm), of Dates, will be taken with breakfast or between breakfast and lunch as a test dose daily (without drinking any tea after it by at least one hour).
  Interventions: Other: Dates fruit as functional Food; Behavioral: behavioral modification and stimulation; Other: nutritional Guidance
- Dates group 2 (Active Comparator): For the group of the date 2, Diagnosed autistic patients matched for age and sex will be given five pieces of Dates will be given on daily basis for 12 weeks as follow: five pieces (each about 10 -15 gm), of Dates, will be taken with breakfast or between breakfast and lunch as a test dose daily (without drinking any tea after it by at least one hour).
  Interventions: Other: Dates fruit as functional Food; Behavioral: behavioral modification and stimulation; Other: nutritional Guidance
- Group 3 (Active Comparator): Group 3 (no- Dates fruit group): Diagnosed autistic patients matched for age and sex will not receive any dates
  Interventions: Behavioral: behavioral modification and stimulation; Other: nutritional Guidance

INTERVENTIONS:
Other: Dates fruit as functional Food — Two groups will receive Dates; The number per group is dependant on the child age. For children aged 3-6 years; they will receive the minimum numbers of dates (3 pieces). For children aged more than 6-12 years will receive 5 pieces of Dates the choice of the minimum numbers of dates (3 pieces) in this current trial is based on a study that was done by Al Jaouni and his colleagues, 2019 which proved the effects of three pieces of Ajwa on infection, hospitalization, and survival among 26 pediatric cancer patients in a university hospital; for which their treatment outcome was improved due to their intake of this amount of Ajwa during their standard treatment
  Arms: Dates group 1; Dates group 2
Behavioral: behavioral modification and stimulation — Behavioral modification applied to the autistic children that is based on applied behavior analysis (ABA), a widely accepted approach that tracks a child's progress in improving his or her skills. We use Positive Behavioral and Support (PBS)
Other: nutritional Guidance — The nutritional education sessions are based on educating parents on providing their autistic children with a nutritious, balanced diet. Because children with ASD often have restricted diets as well as difficulty sitting through meal times, they may not be getting all the nutrients they need, particularly calcium and protein

SUMMARY:
Autism spectrum disorder (ASD) is a lifelong developmental disability that includes deficits in social communication and social interaction and restricted, repetitive patterns of behavior, interests, or activities.

The current treatment approaches for the management of autism are expensive, showing unwanted adverse effects; alter the genetic and metabolic pathways. Many studies referred to the importance of probiotics, minerals and antioxidant supplementation in the treatment of accompanied eating and feeding problems. Meanwhile, there are still controversial results about the effectiveness of dietary interventions for ASD like the gluten-free/casein-free diet and the ketogenic diet.

Dates have been documented in the Holy Quran and proved in modern scientific literature to act as potent antioxidants and as an anti-inflammatory, provide a suitable alternative therapy in various diseases cure.

The medicinal therapeutic value of date fruits as nutritional probiotic and its implications in controlling autism through the anti-oxidant effect will be evaluated. Moreover, at which dose Dates fruit can exert its effect and whether this effect is sustained or not will be also evaluated. Besides, Dates' effect on cognitive, neurological parameters, eating behaviors, and gastrointestinal symptoms and anthropometric measures will be evaluated. A non-randomized clinical study on 120 diagnosed autistic children aged 3-12 years in Cairo will be conducted. Participants will be randomly assigned to one of three groups (each with 40 children) receiving one of three regimens; the first group will receive 3 Dates per day for 3 months and the second group will receive 5 Dates per day for 3 months and the third group will receive nothing. All groups will receive nutrition guidance, behavioral modification, and stimulation sessions. Stools and blood samples will be collected before the study, after 12 weeks of the intervention and then 12 weeks after completion of the intervention. Evaluating Dates' ability to decrease the oxidative stress will be done through comparing blood levels of three oxidative markers; Malondialdehyde (MDA), glutathione peroxidase (GPX1) and superoxide dismutase (SOD) in children with autism for the three proposed regimen. The impact of the Dates fruit consumption on the microbiota of the autistic children both the pathogenic bacteria and probiotics will be done through traditional stool analysis and Real-time PCR before and after interventions.

DETAILED DESCRIPTION:
ASD is progressively increasing; the rate of autism was 3.4 per 1,000 for children aged 3 to 10 years in the 1990s. Meanwhile, in 2006, the prevalence estimates are in the range of 6.5 to 6.6 per 1,000 and recently 1 in 160 children have ASD. Though classified as a neurodevelopmental condition, ASD is often associated with multiple medical comorbidities and gastrointestinal (GI) problems. GI disorders occurred in around 90 % of ASD children with suggested possible role of the GI microflora in the severity of symptoms in autistic children.

Children with ASD frequently have food selectivity, which may have an effect on gastrointestinal symptoms. The gut flora of autistic children is altered compared to healthy children and they have multiple nutritional deficiencies. The microbiota that resides in the gut was claimed to be the cause behind the neurodevelopmental disorders occurring among the autistic children.

Due to the frequent occurrence of gastrointestinal dysfunction in patients with ASD, the use of probiotics may be an indication for adjuvant therapy. Probiotics ''are living nonpathogenic microorganisms, when administered in adequate amounts exert their beneficial effects resulting in modulation of the immune and inflammatory response. The supplementation of probiotic bacteria to autistic children can lead to changes in the microbiota and it considers a useful new therapeutic tool to normalize gut microbiota, restore the function of the epithelial barrier resulting in reliving of the gastrointestinal system disorders, reduce inflammation, and potentially improve the behavioral symptoms in autistic children.

Furthermore, children with autism have deficient antioxidant defense Mechanisms. They are vulnerable to oxidative stress which is detected by elevated lipid peroxidation, especially at younger children. Oxidative stress may play a role in the development and clinical manifestations of autism resulting in loss of acquired language skills in autism. Meguid and coworkers highlighted that autistic children might benefit from antioxidant supplementation coupled with polyunsaturated fatty acids. Early assessment and intervention of antioxidant status may decrease the oxidative stress before inducing more irreversible brain damage.

In Islam, herbs and its constituents have important value in diet and treatment of various types of diseases. The Prophet Mohammed (Peace Be Upon Him) used various herbs and recommended various medicinal plants for the cure of various diseases.

Dates and their constituents show a role in disease prevention through anti-oxidant, anti-inflammatory, anti-bacterial activity. Dates are considered a staple food item in the Middle East and North Africa and are also imported in Europe, the UK, and the USA.

Dates contain relatively high levels of polyphenols and insoluble fiber. It has shown that whole date fruit, and polyphenols extracted from them selectively stimulates Bifidobacterium spp. and Bacteroides, along with the total bacterial counts in fecal batch culture models, increasing small chain fatty acid (SCFA) production concurrently. In addition, promising changes in DNA damage were observed through the anti-proliferative actions of both polyphenol extracts and whole date extracts.

Antioxidant activity of Dates is recognized due to the wide range of phenolic compounds present in Dates including p-coumaric, ferulic, and sinapic acids, flavonoids, and procyanidins.

Dates fruit is considered as a rich source of minerals and sugars; its various constituents like phytochemicals, carotenoids, steroids, and flavonoids are screened for numerous medicine. Rahmani and his colleagues illustrate all the therapeutic functions of the Dates.

Keeping all information in hands about Dates' therapeutic effect in the management of the disease via its anti-oxidant, anti-inflammatory effect and for the sake of autistic children, It is worthy to point and essential to evaluate Dates as a good remedy for autistic children because it is inexpensive and easy to access.

Objectives:

The overall objective is to discover functional food that is effective to control the comorbidities accompanied by autism development and to limit its progression. This food should be safe, inexpensive and affordable, easy to access without any complications.

The medicinal therapeutic value of Dates fruit as nutritional prebiotic and its implications in controlling autism through anti-oxidant and anti-inflammatory effects will be evaluated.

Specific Objectives

The aim of this interventional study is to:

1. Evaluate Dates' effect on cognitive development
2. Evaluate Dates' effect on neurological parameters and severity of autism
3. Evaluate Dates' effect on eating behaviors and diet quality
4. Evaluate Dates' effect on gastrointestinal symptoms and the microbiota
5. Evaluate Dates' ability to decrease the oxidative stress before inducing more irreversible brain damage (through comparing levels of three oxidative markers; Malondialdehyde (MDA), glutathione peroxidase (GPX1) and superoxide dismutase (SOD) in children with autism for the three proposed regimen).
6. Evaluate at which dose Dates fruit can exert its effect as a new therapeutic regimen and its persistence over time

Phases of the study and tools:

This study will be conducted as three phases that will be done in a simultaneous way:

The first phase will include patient recruitment and baseline assessment before Dates fruit intake:

1. Applying the confirmatory diagnostic tools for autistic patients aged 3 -12 years. (Children with suspected ASD could be then assessed according to either Diagnostic and statistical manual of mental disorders, 5th edition. (DSM-V) criteria, and CARS.

An autism screening tool must meet all three primary areas defined by the DSM-V description for the autistic disorder to qualify for a positive rating from First Signs:

A. A total of six (or more) items from (1), (2), and (3), with at least two from (1), and one each from (2) and (3):

1. Qualitative impairment in social interaction, as manifested by at least two of the following:

   1. Marked impairment in the use of multiple nonverbal behaviors, such as eye-to-eye gaze, facial expression, body postures, and gestures to regulate social interaction
   2. Failure to develop peer relationships appropriate to the developmental level
   3. A lack of spontaneous seeking to share enjoyment, interests, or achievements with other people (e.g., by a lack of showing, bringing, or pointing out objects of interest)
   4. Lack of social or emotional reciprocity
2. Qualitative impairments in communication, as manifested by at least one of the following:

   1. Delay in, or total lack of, the development of spoken language (not accompanied by an attempt to compensate through alternative modes of communication such as gesture or mime)
   2. In individuals with adequate speech, marked impairment in the ability to initiate or sustain a conversation with others
   3. Stereotyped and repetitive use of language or idiosyncratic language
   4. Lack of varied, spontaneous make-believe play or social imitative play
3. Restricted, repetitive, and stereotyped patterns of behavior, interests, and activities as manifested by at least one of the following:

   1. Encompassing preoccupation with one or more stereotyped and restricted patterns of interest that is abnormal either in intensity or focus
   2. Apparently inflexible adherence to specific, nonfunctional routines or rituals
   3. Stereotyped and repetitive motor mannerisms (e.g., hand or finger flapping or twisting or complex whole-body movements)
   4. Persistent pre-co-occupation with parts of objects B. Delays or abnormal functioning in at least one of the following areas, with onset prior to age 3 years: (1) social interaction, (2) language as used in social communication, or (3) symbolic or imaginative play.

      The Instruments of the investigation will also include socio-demographic assessment questionnaire including suggested history of risk factors (Demographics, Medication exposure, Medical conditions, Pesticides, Diet, Home environmental exposures, Health behaviors/lifestyle, Mental condition/history/symptoms, Vaccine history, Personal product use, Anthropometrics, Medical procedures, Occupational history. In addition, the questionnaire will focus on socioeconomic indicators as well as prenatal and perinatal and neonatal risk factors such as the timing of conception, weight gain during pregnancy, parental age, and inter-pregnancy interval.

      2. Assessment of the sociodemographic characteristics through detailed history taking, pregnancy history, peri-natal history, and other risk factors

      3. Neurological assessment through thorough clinical examination

      4. Assessing functional gastrointestinal behavior disorders (FGID): Assessing changes in the GI symptoms which may be constipation, diarrhea, gaseousness, bloating, gastroesophageal reflux, abdominal pain, and vomiting but constipation is the more common and the most reported GI symptoms

      5. Detailed nutritional and dietary assessment with anthropometric measurements Anthropometric measurements
      1. Weight (in kg): by Body fat analyzer
      2. Height (in cm): using Stadiometer
      3. BMI (weight/Height2 in meter):calculated
      4. Waist circumference (in cm): measuring tapes
      5. Hip circumference (in cm): measuring tapes
      6. Waist / Hip ratio: calculated
      7. measuring body composition analyzer (Bioelectrical impedance) for autistic children aged seven years and older (measure fat mass, fat-free mass, fat %, water content, Basal metabolic rate (BMR)

      6. Behavioral Assessment; the interview questions will cover eight content areas:
      1. The subject's background, including family, education, previous diagnoses, and medications
      2. Overview of the subject's behavior
      3. Early development and developmental milestones
      4. Language acquisition and loss of language or other skills
      5. Current functioning in regard to language and communication
      6. Social development and play
      7. Interests and behaviors
      8. Clinically relevant behaviors, such as aggression, self-injury, and possible epileptic features

      Mental Development, Psychomotor Development and Behavior Rating will be assessed by using the "Bailey Scales of Infant and Toddler Development", the cognitive, language, and motor abilities will be assessed; as well as social-emotional and adaptive behavior. Mental and psychomotor developmental quotients and mental age will be scored as well as the behavioral profile. The Bailey Screening Test is an Observation Checklist for 5 domains of development (cognitive, language, motor, social-emotional, & adaptive behavior).

      The questionnaire will be directed for the mothers of all confirmed cases with ASD enrolled in the study

      Second phase Intervention phase

      Special emphasis will be directed towards focusing on treating accompanied neurological manifestations Third phase: during this phase, the outcome of the intervention on the stool microbiota and on the serum antioxidant markers will be evaluated twice; once after completing the intervention and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Is not allergic to Dates (tested initially by one piece of Dates)
* Agrees to the intake of Dates fruits for at least 3 months
* Not participating in another study
* Signed the consent to participate in the study
* Caregiver consent was obtained for all the studied cases.

Exclusion Criteria:

* All subjects with other causes of mental sub-normality and/or delayed language
* Refuses intake of Dates
* Participating in another study
* Refused to sign the consent to participate in the study
* Patients who consumed probiotics and/or Dates for at least 4 weeks prior to the trial and/or antibiotics or laxatives for 6 months prior to the start.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Dates' ability to change the oxidative stress of ASD | ifference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  comparing blood levels of three oxidative markers; Malondialdehyde (MDA), glutathione peroxidase (GPX1) and superoxide dismutase (SOD) in children with autism for the three proposed regimen. Measuring the difference pre and three months after the intervention, before and six months after the intervention
change on the pathogenic microbiota of the autistic children as detected by traditional stool analysis through DNA extraction (quantitative PCR) of the fecal samples | ifference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  Through the quantitative PCR (qPCR) for the change in the presence and absence of the targeted bacterial subgroups (including Bifidobacterium, lactobacillus, Clostridium, Sutterella)
change on the useful microbiota of the autistic children ( probiotics) | ifference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  by DNA extraction kits of the fecal samples and Real-time PCR before and after interventions we will measure the change in the presence of the probiotics before and after the intervention

SECONDARY OUTCOMES:
Dates' effect on the change of the behavioral rating assessed by an Observation Checklist using the "Bailey Scales of Infant and Toddler Development | The difference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  Mental Development, Psychomotor Development and Behavior Rating will be assessed by using the "Bailey Scales of Infant and Toddler Development", the cognitive, language, and motor abilities will be assessed; as well as social-emotional and adaptive behavior. Mental and psychomotor developmental quotients and mental age will be scored as well as the behavioral profile. The Bailey Screening Test is an Observation Checklist for 5 domains of development (cognitive, language, motor, social-emotional, & adaptive behavior).
Dates' effect on the change of the mental development assessed by an Observation Checklist using the "Bailey Scales of Infant and Toddler Development" | The difference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  Mental Development, Psychomotor Development and Behavior Rating will be assessed by using the "Bailey Scales of Infant and Toddler Development", the cognitive, language, and motor abilities will be assessed; as well as social-emotional and adaptive behavior. Mental and psychomotor developmental quotients and mental age will be scored as well as the behavioral profile. The Bailey Screening Test is an Observation Checklist for 5 domains of development (cognitive, language, motor, social-emotional, & adaptive behavior).
Dates' effect on the change of the Psychomotor abilities assessed by the observational checklist using the "Bailey Scales of Infant and Toddler Development | The difference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  Mental Development, Psychomotor Development and Behavior Rating will be assessed by using the "Bailey Scales of Infant and Toddler Development", the cognitive, language, and motor abilities will be assessed; as well as social-emotional and adaptive behavior. Mental and psychomotor developmental quotients and mental age will be scored as well as the behavioral profile. The Bailey Screening Test is an Observation Checklist for 5 domains of development (cognitive, language, motor, social-emotional, & adaptive behavior).
Dates' effect on the changes of the level of the autism as assessed by the 5th edition of the DSM-V | The difference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  comparing changes the severity of autism as a result of interventions according Diagnostic and statistical manual of mental disorders, 5th ed. (DSM-V) criteria it measure specific ASD symptom severity All core features of ASD are included: socialisation impairments, communication deficits and repetitive or restricted interests, including sensory abnormalities. After a period of interactive play, the observer rates the child's behaviour, comparing it to that of his/her age group. Each item is given a numerical score of '0' (indicating no impairment), '1' (indicating mild impairment), or '2' (indicating severe impairment)
Dates' effect on the changes of the severity of the autism as assessed by Childhood Autism Rating Scale (CARS) measure | The difference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  comparing changes the severity of autism as a result of interventions according to CARS.Each item on the Clinician-Rated Severity of Autism Spectrum and Social Communication Disorders measure is rated on a 4-point scale (Level 0=None; Level 1=Mild/Requiring support; Level 2=Moderate/Requiring SUBSTANTIAL support; and Level 3=Severe/Requiring VERY SUBSTANTIAL support).
Dates' effect on the change on the dietary intake using the Food frequency questionnaire, 24-hour dietary recall, Dietary record | The difference from the initial (before the intervention) with that three and Six months after the initiation of the intervention
  comparing changes on eating behaviors as assessed by the 24 hours intake and food pattern. Dietary intake is difficult to measure, and any single method cannot assess dietary exposure perfectly. The 24HR, and FFQ are subjective estimates. Recently, it has been suggested that a combination of methods, such as the FFQ with 24HR be used to obtain more accurate estimates of dietary intakes than that of individual methods. They are widely used as the primary dietary assessment tool in epidemiological studies..

CONTACTS AND LOCATIONS:
Overall Officials: Ammal M Metwally, PhD, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after the end of the project
Access Criteria: the data will be accessed through a drive with a link

REFERENCES:
- [Background] 1- World Health Organization (WHO). Autism Spectrum Disorders, Fact sheet, https://www.who.int/news-room/fact-sheets/detail/autism-spectrum-disorders, acessesd on 1-7-2019, 2018
- [Background] Kohane IS, McMurry A, Weber G, MacFadden D, Rappaport L, Kunkel L, Bickel J, Wattanasin N, Spence S, Murphy S, Churchill S. The co-morbidity burden of children and young adults with autism spectrum disorders. PLoS One. 2012;7(4):e33224. doi: 10.1371/journal.pone.0033224. Epub 2012 Apr 12. PMID 22511918
- [Background] McElhanon BO, McCracken C, Karpen S, Sharp WG. Gastrointestinal symptoms in autism spectrum disorder: a meta-analysis. Pediatrics. 2014 May;133(5):872-83. doi: 10.1542/peds.2013-3995. PMID 24777214
- [Background] Kushak R., Buie T.: Intestinal disaccharidase deficiency in children with autism spectrum disorders. J. Pediatr. Gastroent. 2002; 35,:436.
- [Background] Israelyan N, Margolis KG. Reprint of: Serotonin as a link between the gut-brain-microbiome axis in autism spectrum disorders. Pharmacol Res. 2019 Feb;140:115-120. doi: 10.1016/j.phrs.2018.12.023. Epub 2019 Jan 15. PMID 30658882
- [Background] Li Q, Zhou JM. The microbiota-gut-brain axis and its potential therapeutic role in autism spectrum disorder. Neuroscience. 2016 Jun 2;324:131-9. doi: 10.1016/j.neuroscience.2016.03.013. Epub 2016 Mar 8. PMID 26964681
- [Background] Meguid NA, Dardir AA, Abdel-Raouf ER, Hashish A. Evaluation of oxidative stress in autism: defective antioxidant enzymes and increased lipid peroxidation. Biol Trace Elem Res. 2011 Oct;143(1):58-65. doi: 10.1007/s12011-010-8840-9. Epub 2010 Sep 16. PMID 20845086
- [Background] Perry G, Nunomura A, Harris S, Smith M, Salomon R., Is Autism a disease of oxidative stress.Oxidative stress in autism symposium, New York State, Institute for basic research in Developmental Disabilities. 2005; p. 15
- [Background] Gebril OH, Meguid NA. HFE gene polymorphisms and the risk for autism in Egyptian children and impact on the effect of oxidative stress. Dis Markers. 2011;31(5):289-94. doi: 10.3233/DMA-2011-0830. PMID 22048270
- [Background] Dar-ul-Iman Healing,. Food of the Prophet (Sallallaho Alayhi Wasallam) Available at: http://chishti.org/foods_of_the_prophet. acessesd on 1-7-2019, 2000
- [Background] Marwat SK, Khan MA, Rehman F, Bhatti IU. Aromatic plant species mentioned in the Holy Qura'n and Ahadith and their ethnomedicinal importance. Pak J Nut. 2009;8: 1472-1479.
- [Background] Eid N, Enani S, Walton G, Corona G, Costabile A, Gibson G, Rowland I, Spencer JP. The impact of date palm fruits and their component polyphenols, on gut microbial ecology, bacterial metabolites and colon cancer cell proliferation. J Nutr Sci. 2014 Oct 8;3:e46. doi: 10.1017/jns.2014.16. eCollection 2014. PMID 26101614
- [Background] Mansouri A, Embarek G, Kokkalou E, Kefalas P. Phenolic profile and antioxidant activity of the Algerian ripe date palm fruit (Phoenix dactylifera) Food Chem. 2005;89:411-420.
- [Background] Gu L, Kelm MA, Hammerstone JF, Beecher G, Holden J, Haytowitz D, Prior RL. Screening of foods containing proanthocyanidins and their structural characterization using LC-MS/MS and thiolytic degradation. J Agric Food Chem. 2003 Dec 3;51(25):7513-21. doi: 10.1021/jf034815d. PMID 14640607
- [Background] Mirza MB, Syed FQ, Khan F, Elkady AI, Al-Attar AM, Hakeem KR. Ajwa Dates: A Highly Nutritive Fruit with the Impending Therapeutic Application. In: Plant and Human Health, Volume 3. Cham: Springer International Publishing; 2019;. 209-30.
- [Background] Sheikh BY, Zihad SM, Sifat N, Uddin SJ, Shilpi JA, Hamdi OA, Hossain H, Rouf R, Jahan IA. Comparative study of neuropharmacological, analgesic properties and phenolic profile of Ajwah, Safawy and Sukkari cultivars of date palm (Phoenix dactylifera). Orient Pharm Exp Med. 2016;16(3):175-183. doi: 10.1007/s13596-016-0239-5. Epub 2016 Aug 16. PMID 27746708
- [Background] Rahmani AH, Aly SM, Ali H, Babiker AY, Srikar S, Khan AA. Therapeutic effects of date fruits (Phoenix dactylifera) in the prevention of diseases via modulation of anti-inflammatory, anti-oxidant and anti-tumour activity. Int J Clin Exp Med. 2014 Mar 15;7(3):483-91. eCollection 2014. PMID 24753740